CLINICAL TRIAL: NCT07216872
Title: A Prospective, Double Blind, Randomized, Controlled Study to Evaluate the Safety and Effectiveness of the BrainsWay Deep Transcranial Magnetic Stimulation (Deep TMS) for Treatment of Alcohol Use Disorder (AUD)
Brief Title: Safety and Effectiveness of the BrainsWay Deep Transcranial Magnetic Stimulation (Deep TMS) for Treatment of Alcohol Use Disorder (AUD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTP-AUD-00
Record Dates: First submitted 2025-10-12; First posted 2025-10-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Alcoholism; Alcohol Abuse; Alcohol Dependence; Alcohol Abuse/Dependence; Alcohol Addiction
Keywords: alcohol use disorder; alcoholism; alcohol abuse; alcohol dependence; alcohol addiction; DTMS; rfTMS; Brainsway
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, sham-controlled, multicenter trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment group (Experimental): The treatment group will receive active, Deep TMS treatment.
  Interventions: Device: Deep TMS (DTMS)
- Control group (Sham Comparator): The Control group will receive inactive, sham treatment.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Deep TMS (DTMS) — The Deep TMS group will receive 30 active sessions in 15 visits (i.e., 2 treatments per visit) over a period of 3-5 weeks in the Acute Treatment Phase. In the Maintenance Treatment & Follow-up phase subjects will receive one treatment session per week from the end of the Acute Treatment Phase until the 6-month follow-up visit. All treatment sessions will consist of 2 treatments per day with a 30 minute interval in between. Each treatment will last approximately 20 minutes.
  Arms: Treatment group
Device: Sham (No Treatment) — The control group will receive 30 Sham sessions in 15 visits (i.e., 2 treatments per visit) over a period of 3-5 weeks in the Acute Treatment Phase. In the Maintenance Treatment & Follow-up phase subjects will receive one treatment session per week from the end of the Acute Treatment Phase until the 6-month follow-up visit. All treatment sessions will consist of 2 treatments per day with a 30 minute interval in between. The control group will receive inactive/sham treatment with identical parameters to the Deep TMS treatment.
  Arms: Control group

SUMMARY:
The study will compare alcohol use in two groups of subjects. One group will be assigned to the Deep TMS treatment and the other group will be assigned to the sham treatment. This is a prospective, 6-month, double blind, randomized, controlled, multi-center trial in outpatients recruited in both academic and private research centers. The study population will consist of subjects diagnosed with moderate to severe AUD. The study is comprised of three phases:

1. Pre-study Screening and Baseline Phase
2. Acute Treatment Phase and
3. Maintenance Treatment and Follow up Phase

Subjects of all ethnic and gender categories, ages ranging between 18-86 years will be screened for study eligibility according to the inclusion and exclusion criteria. Subjects who meet the eligibility criteria and are willing to sign an informed consent form will be enrolled in the study. The subjects' demographic and baseline characteristics, as well as their overall medical condition will be assessed prior to treatment administration.

Eligible patients will be randomized with a 1:1 ratio to one of two study groups (treatment or sham) and stratified by site. Randomization will be employed to avoid bias in the assignment of subjects to treatment group. All subjects will undergo the same treatment regimen, regardless of the assigned treatment group. The acute treatment phase will include 15 treatment visits over a period of 3-5 weeks.

The Maintenance Treatment & Follow-up phase will include one treatment visit per week from the end of the Acute Treatment Phase until the 6 month follow-up visit.

At each treatment session, prior to stimulation onset, alcohol related cues will be presented to the subject. After the offset of the alcohol cue presentation, active or sham Deep TMS stimulation will be administered.

The study design is directed towards a comparison between active treatment and sham, up to 4 months and 6 months follow-up. Efficacy will be assessed using the primary efficacy measure of the percent heavy drinking days during months 2-4, based on the Time Line Follow Back (TLFB) reporting. Additionally, several subject assessment scales will be used during the course of the study to assess alcohol use and alcohol craving.

Safety will be assessed, including monitoring the severity, causality and frequency of all adverse events, vital signs, and physical and neurological examination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-86 years old.
2. Subjects diagnosed with AUD and who meet criteria for moderate (4-5 out of the 12 symptoms) to severe (> 6 out of the 12 symptoms) AUD according to the DSM-5 diagnostic criteria as determined by a licensed clinician according to the DSM-5 criteria, and verified with the Mini International Neuropsychiatric Interview (Standard MINI version 7.0.2).
3. Subjects who have a history of at least 24 heavy drinking days during the 90 days prior to screening (average >=8 HDD/month), based on TLFB).
4. Treatment seeking individuals with a treatment goal of achieving abstinence or reducing heavy drinking.
5. Subjects able to understand and provide signed informed consent, and able to adhere to the requirements and restrictions of this protocol.
6. Satisfactory answers on safety screening questionnaire for transcranial magnetic stimulation.

Exclusion Criteria:

1. Subjects diagnosed with schizophrenia or chronic psychotic disorder as determined by a licensed clinician according to the DSM-5 criteria, and verified with the Mini International Neuropsychiatric Interview (Standard MINI version 7.0.2).
2. Subjects with present suicidal risk as assessed by the investigator or significant suicide risk based on MADRS item 10 score of 4 or 6, or a history of attempted suicide in the last year.
3. Subjects who initiated treatment with any of the following medications which are known to effect alcohol consumption, within 30 days of the Screening visit: acamprosate, baclofen, buprenorphine, disulfiram, gabapentin, naltrexone, topiramate and varenicline.
4. Subjects with a significant medical illness that is not well controlled (e.g., hepatic impairment, diabetes, hypertension, heart disease, septicemia, active tuberculosis, progressive neoplasm, frequent and severe migraine headaches, etc.).
5. Subjects experiencing acute alcohol withdrawal. This will be determined using the Clinical Institute Withdrawal Assessment of Alcohol - revised (CIWA-Ar) wherein subjects with a value of >7 will not be permitted to receive TMS on that day to mitigate any potential risk of a seizure. Treatments may be rescheduled and CIWA-AR and alcohol breath tests may be reassessed, although if more than the allowed treatment sessions are missed, the subject will be withdrawn from the study.
6. Subjects with a history of epilepsy or seizure (not including history of alcohol withdrawal seizure, ECT induced seizures, or childhood febrile seizures).
7. Individuals with a first-degree relative family history of seizure.
8. Subjects with a high risk for severe violence or suicidality as assessed during the screening interview.
9. Conductive, ferromagnetic or other magnetic-sensitive metals implanted in the head (outside the mouth) or within 10 cm of the treatment coil (e.g., cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, shrapnel, surgical clips, fragments from welding or metal work).
10. Subjects with cardiac pacemakers or active implantable electrodes/neurostimulators within 30 cm of the treatment coil.
11. Subjects with a significant neurological disorder or insult including, but not limited to:

    * Any condition likely to be associated with increased intracranial pressure
    * Space occupying brain lesion
    * History of cerebrovascular accident
    * Transient ischemic attack within two years
    * Cerebral aneurysm
    * Dementia
    * Mini Mental State Exam score of less than or equal to 24
    * Parkinson's disease
    * Huntington's chorea
    * Multiple sclerosis
12. Subjects suffering from significant hearing loss.
13. Previous treatment with TMS within one year.
14. Participation in another clinical investigation in which a device or drug has been used within 4 weeks of screening.
15. If participating in psychotherapy, subject is not in stable treatment for at least 3 months prior to entry into the study or anticipates a change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial.
16. Known or suspected pregnancy or lactation or planning to become pregnant.
17. Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of patients who attain zero (0) heavy drinking days | 2-4 months
  The difference in the proportion of patients who attain zero (0) heavy drinking days in the Treatment group versus the Sham control group in months 2-4 following initiation of the Acute Phase, based on TLFB reporting. Month 1 is considered a "Grace Period" as this is the time during which the full treatment dose of the Acute Phase is being delivered.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Alpha Neuron LLC, Tuscaloosa, Alabama
  - Kadima Neuropsychiatry, La Jolla, California
  - DTMS Center LLC, West Palm Beach, Florida
  - Rosecrance River North, Chicago, Illinois
  - ManuMind Interventional Psychiatry, Woodbury, New York
  - PsyCare, South Charleston, West Virginia
- Soroka Medical Center, Beersheba, Israel